CLINICAL TRIAL: NCT03190304
Title: The Effect of NEPRIlysin (LCZ696) on EXercise TOLerance, Muscle Vasodilatation, Muscle Strength and Body Composition in Patients With Heart Failure - NEPRIExTol-HF Trial
Brief Title: The Effect of Neprilysin (LCZ696) on Exercise Tolerance in Patients With Heart Failure
Acronym: NEPRIExTol
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NEPRIExTol-HF Trial
Record Dates: First submitted 2017-06-14; First posted 2017-06-16 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-03

CONDITIONS: Heart Failure; Exercise Tolerance; Vasodilation; Body Composition; Muscle Strength
MeSH Terms: conditions — Heart Failure; Aneurysm | interventions — Neprilysin; sacubitril and valsartan sodium hydrate drug combination; Enalapril; Angiotensin-Converting Enzyme Inhibitors

STUDY DESIGN:
Intervention Model Description: double-blind, randomized clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Enalapril (Active Comparator): Enalapril at a dose of 10 mg twice daily for 6 months
  Interventions: Drug: Enalapril
- Neprilysin (LCZ696) (Experimental): LCZ696 at a dose of 200 mg twice daily for 6 months
  Interventions: Drug: Neprilysin

INTERVENTIONS:
Drug: Neprilysin — To compare the effect of Enalapril and Neprilysin on exercise tolerance in patients with heart failure
  Other Names: LCZ696
  Arms: Neprilysin (LCZ696)
Drug: Enalapril — To compare the effect of Enalapril and Neprilysin on exercise tolerance in patients with heart failure
  Other Names: Angiotensin converting enzyme inhibitor
  Arms: Enalapril

SUMMARY:
Studies with new drugs in the treatment of heart failure (HF), such as the combination of valsartan/sacubitril, also known as LCZ696, have demonstrated important clinical impact on the morbidity and mortality outcomes in HF population. However, the effect of LCZ696 on the pathophysiological mechanisms of HF such as exercise tolerance (peak VO2) and peripheral muscle blood flow is not known. Since LCZ696 is a new drug with promising effects on the treatment of HF, the objective of the present study will be to evaluate the effect of LCZ696 in patients with HF on: 1) peak VO2, 2) 6-minute walk test, 3) peripheral muscle blood flow, 4) muscle strength, and 5) body composition.

DETAILED DESCRIPTION:
Heart failure (HF) with reduced ventricular ejection fraction is a disease that affects around 5.7 million people in the United States, with a mortality rate of approximately 50% within 5 years. HF is characterized by an exacerbation of the renin-angiotensin-aldosterone system (RAAS), which leads to an increase in sympathetic nerve outflow, peripheral vasoconstriction, and reduced functional capacity. Moreover, many clinical trials have been developed for the treatment of HF patients focused on inhibition of RAAS, such as enalapril. Nevertheless, hospitalization and mortality rates in this population are excessive. However, studies with new drugs, such as the combination of valsartan/sacubitril, also known as LCZ696, have demonstrated important clinical impact on the morbidity and mortality outcomes in HF population. However, the effect of LCZ696 on the pathophysiological mechanisms of HF such as exercise tolerance (peak VO2) and peripheral muscle blood flow is not known. Since LCZ696 is a new drug with promising effects on the treatment of HF, the objective of the present study will be to evaluate the effect of LCZ696 in patients with HF on: 1) peak VO2, 2) 6-minute walk test, 3) peripheral muscle blood flow, 4) muscle strength, and 5) body composition.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic patients with heart failure (men and women) aged >18 years,
2. Functional class II, III or IV by the New York Heart Association (NYHA)
3. Left ventricular ejection fraction <35%
4. Ischemic and nonischemic etiology
5. Type B natriuretic peptide (BNP) >150 pg/ml (or pro-BNP [N-terminal-proBNP] ≥ 600 pg / ml) or if the patient was hospitalized for cardiac decompensation within the preceding 12 months, BNP >100 pg/ml (or N-terminal-proBNP ≥ 400 pg / ml)

Exclusion Criteria:

1. History of hypersensitivity or allergy to any of the study drugs, drugs of similar chemical classes, ACE inhibitors (ACEIs), angiotensin II receptor blockers (ARBs), or neprilysin inhibitors, as well as known or suspected contraindications to the study drugs.
2. Previous history of intolerance to recommended target doses of ACEIs or ARBs.
3. Known history of angioedema.
4. Requirement for treatment with both ACEIs and ARBs.
5. Current acute decompensated heart failure (exacerbation of chronic heart failure manifested by signs and symptoms that may require intravenous therapy).
6. Symptomatic hypotension.
7. Estimated glomerular filtration rate (eGFR) <30%.
8. Serum potassium >5.4 mmol/L.
9. Acute coronary syndrome, stroke, transient ischaemic attack, cardiac, carotid, or other major cardiovascular surgery, percutaneous coronary intervention, or carotid angioplasty within the 3 months.
10. Coronary or carotid artery disease likely to require surgical or percutaneous intervention within the 6 months.
11. Implantation of a cardiac resynchronization therapy (CRT) device within 3 months or intent to implant a CRT.
12. History of heart transplant or on a transplant list or with left ventricular (LV) assistance device.
13. History of severe pulmonary disease.
14. Diagnosis of peripartum- or chemotherapy-induced cardiomyopathy within the 12 months.
15. Documented untreated ventricular arrhythmia with syncopal episodes within the 3 months.
16. Symptomatic bradycardia or second- or third-degree atrioventricular block without a pacemaker.
17. Presence of haemodynamically significant mitral and/or aortic valve disease, except mitral regurgitation secondary to LV dilatation.
18. Presence of other haemodynamically significant obstructive lesions of the LV outflow tract, including aortic and subaortic stenosis.
19. Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of study drugs, including, but not limited to, any of the following: History of active inflammatory bowel disease during the 12 months. Active duodenal or gastric ulcers during the 3 months. Evidence of hepatic disease as determined by any one of the following: aspartate aminotransferase or alanine aminotransferase values exceeding 2x upper limit of normal, history of hepatic encephalopathy, history of oesophageal varices, or history of porto-caval shunt. Current treatment with cholestyramine or colestipol resins.
20. Presence of any other disease with a life expectancy of <5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2020-09-14 (Actual); Study Completion 2020-09-23 (Actual)

PRIMARY OUTCOMES:
Exercise tolerance | 6 months
  To test the effect of treatments on peak oxygen consumption

SECONDARY OUTCOMES:
Walking distance | 6 months
  To test the effect of treatments on 6 minutes walking test
Muscle vasodilation | 6 months
  To test the effect of treatments on forearm blood flow evaluated by venous occlusion plethysmography
Muscle strength | 6 months
  To test the effect of treatments on muscle strength evaluated by handgrip
Body composition | 6 months
  To test the effect of treatments on lean muscle mass evaluated by dual energy x-ray absorptiometry

CONTACTS AND LOCATIONS:
Overall Officials: Antonio P Barretto, PhD, Principal Investigator — Heart Institute (InCor), University of Sao Paulo Medical School
Locations (1):
- Marcelo Rodrigues dos Santos, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dos Santos MR, Alves MNN, Jordao CP, Pinto CEN, Correa KTS, de Souza FR, da Fonseca GWP, Tomaz Filho J, Costa M, Pereira RMR, Negrao CE, Barretto ACP. Sacubitril/valsartan versus enalapril on exercise capacity in patients with heart failure with reduced ejection fraction: A randomized, double-blind, active-controlled study. Am Heart J. 2021 Sep;239:1-10. doi: 10.1016/j.ahj.2021.05.005. Epub 2021 May 14. PMID 33992607